CLINICAL TRIAL: NCT02551250
Title: Comparison of Biannual Ultrasonography and Annual Unenhanced Magnetic Resonance Imaging as a Surveillance Test for Hepatocellular Carcinoma in Patients With Liver Cirrhosis
Brief Title: Annual MRI Versus Biannual US for Surveillance of Hepatocellular Carcinoma in Liver Cirrhosis
Acronym: MAGNUS-HCC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: JOON-IL CHOI (Other)
Collaborators: Seoul National University Hospital (Other); Samsung Medical Center (Other); Korea University Guro Hospital (Other); The Catholic University of Korea (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor-Investigator, JOON-IL CHOI, Associate professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: 1520160
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Liver Cirrhosis
Keywords: hepatocellular carcinoma; surveillance; liver cirrhosis; ultrasonography; magnetic resonance imaging
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study: Surveillance of HCC by biannual ultrasonography AND annual noncontrast MRI
  Interventions: Device: annual noncontrast MRI; Device: biannual ultrasonography

INTERVENTIONS:
Device: annual noncontrast MRI — liver MRI without contrast agents T2 weighted image, T1 in/out of phase, diffusion weighted images with b-values of 0, 500 mm2/s
Device: biannual ultrasonography — liver ultrasonography for HCC screening performed by experienced sonologists

SUMMARY:
The investigators will investigate the usefulness of biannual ultrasonography versus annual non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma in single arm patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the major complications in patients with chronic liver disease. The prognosis of HCC relies on the extent of disease at the time of diagnosis. Hence to detect cancer at an earlier stage, a regular surveillance test is important for the subjects with a high risk of developing cancer. Current guidelines recommend a regular surveillance using ultrasonography (US) at a 6 month-interval. Ultrasonography is a non-invasive and safe procedure, yet it is limited by the skills of the operator and it is often difficult to differentiate cancer from regenerating nodules especially in atrophied cirrhotic liver. According to a recent meta-analysis, the overall sensitivity and specificity of detecting liver cancer using ultrasonography were both over 90%, however the sensitivity was decreased to 60% in detecting early lesions in which surgery or liver transplantation is indicated. Of note, addition of alpha feto protein(AFP) to ultrasonography also failed to increase the sensitivity in detecting small cancers. Taken together, there is a need to develop a new surveillance test with an improved sensitivity and specificity.

Recently, a retrospective study reported that CT or MRI showed a better sensitivity than ultrasonography in detecting early liver cancer. However, performing CT as a surveillance test is limited by frequent exposure to radiation and contrast-dye agent. Although MRI does not have the risk of radiation-exposure, it is limited by the high cost and limited availability. On the contrast, non-contrast MRI offers a cost that is comparable to US and an absence of exposure to radiation or contrast-dye agent, which suggests non-contrast MRI as a good alternative surveillance tool for early detection of HCC. Therefore, in this prospective trial, the investigators will investigate the usefulness of biannual ultrasonography versus annual non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject older than 40 years of age at the enrollment
* Fulfill below conditions A and B

A. The evidence of cirrhosis of any etiology within 12 months prior to screening Definition of cirrhosis by any of following methods

1. Histologically by liver biopsy;
2. Non-histologically by evidence of portal hypertension in the presence of chronic liver disease;

   * Evidence of portal hypertension, including any of followings;

     * The identification of splenomegaly on ultrasonography, CT, or MRI examinations with typical features of cirrhosis
     * The identification of esophageal or gastric varices on endoscopic examination

B. Risk Index larger than 2.33; Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100,000/mm3) + 0.74 (if the presence of HCV is positive).

Exclusion Criteria:

* Presence of liver cancer or other intrahepatic malignancy
* Has a history of malignancy within previous 5 years
* Is pregnant or breast-feeding

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the risk of annual HCC occurrence larger than 5%
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity for detecting HCC | 3 years
  sensitivity for detecting HCC

SECONDARY OUTCOMES:
survival of the patients who developed HCC on follow-up period | years
  survival of the patients who developed HCC on follow-up period
false referral rate for HCC | 3 years
  false referral rate for HCC

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Il Choi, Principal Investigator — Seoul St. Mary's Hospital
Locations (6):
- South Korea (6):
  - Seoul St.Mary's Hospital, Seoul
  - Korean University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - St.Vincent's Hospital, Suwon
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim YK, Kim YK, Park HJ, Park MJ, Lee WJ, Choi D. Noncontrast MRI with diffusion-weighted imaging as the sole imaging modality for detecting liver malignancy in patients with high risk for hepatocellular carcinoma. Magn Reson Imaging. 2014 Jul;32(6):610-8. doi: 10.1016/j.mri.2013.12.021. Epub 2014 Jan 13. PMID 24702980
- [Derived] Kim DH, Yoon JH, Choi MH, Lee CH, Kang TW, Kim HA, Ku YM, Lee JM, Kim SH, Kim KA, Lee SL, Choi JI. Comparison of non-contrast abbreviated MRI and ultrasound as surveillance modalities for HCC. J Hepatol. 2024 Sep;81(3):461-470. doi: 10.1016/j.jhep.2024.03.048. Epub 2024 Apr 16. PMID 38636849
- [Derived] Kim HA, Kim KA, Choi JI, Lee JM, Lee CH, Kang TW, Ku YM, Lee SL, Park YS, Yoon JH, Kim SH, Choi MH. Comparison of biannual ultrasonography and annual non-contrast liver magnetic resonance imaging as surveillance tools for hepatocellular carcinoma in patients with liver cirrhosis (MAGNUS-HCC): a study protocol. BMC Cancer. 2017 Dec 21;17(1):877. doi: 10.1186/s12885-017-3819-y. PMID 29268722